CLINICAL TRIAL: NCT05847803
Title: Nurses' Perceptions of Patient Monitoring in the Intensive Care Unit: a Cross-sectional Study
Brief Title: Patient Monitoring in the Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20230110
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-01

CONDITIONS: Medical Informatics; Intensive Care

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, questionnaire survey — No intervention, questionnaire survey

SUMMARY:
a cross-sectional survey of nurses' perception of patient monitoring in the ICUs

ELIGIBILITY:
Inclusion Criteria:

* registered nurses in the ICUs

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: registered nurses in the ICUs
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
clinical requirements of patient monitoring in ICUs | 12 months of working
  Assessed using a web-based 36-item survey questionnaire Patient Monitoring in the Intensive Care Unit
Work-related flow in ICUs | 12 months of working
  Assessed using the Work-related Flow inventory (WOLF)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Gao, PhD, Study Chair — SAHZU
Locations (1):
- SAHZhejiangU, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No